CLINICAL TRIAL: NCT04198064
Title: Pain Management for Cystoscopy: A Prospective Randomized Study Focused on Understanding the Role of the "Bag Squeeze" to Manage Pain for Patients Undergoing Cystoscopy
Acronym: PMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19-5661
Record Dates: First submitted 2019-10-01; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Pain, Procedural
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A- Bag Squeeze (Experimental): Participants will receive a "bag squeeze" of irrigation fluid (500 ml/~2 cups of %0.9 saline solution) during the insertion of the cystocopy tube during their cystoscopy.
  Interventions: Procedure: Bag Squeeze
- Group B- No Bag Squeeze (Other): Participants will receive a standard cystoscopy procedure.
  Interventions: Procedure: No Bag Squeeze

INTERVENTIONS:
Procedure: Bag Squeeze — Participants will receive a "bag squeeze" of irrigation fluid (500 ml/~2 cups of % 0.9 saline solution) during the insertion of the cystocopy tube during their cystocopy.
  Arms: Group A- Bag Squeeze
Procedure: No Bag Squeeze — Participants will receive a standard cystocopy procedure as per standard of care.
  Arms: Group B- No Bag Squeeze

SUMMARY:
The purpose of this study is to determine whether utilization of the "bag squeeze" technique during flexible cystoscopy changes pain scores using a study questionnaire designed by the team which comprises a validated Lingard pain rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Undergoing flexible cystocopy at University Health Network that have undergone a flexible cystocopy and did not demonstrate difficulty during exploration (meatal stenosis or urethral stricture), simultaneous removal or ureteral stents or bladder biopsies or have a chronic history of pelvic pain

Exclusion Criteria:

- Patients that do not meet the inclusion criteria.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Pain Rating | The outcome measure will be assessed for up to 4 hours after consent and completion of clinical procedure.
  Participants will be asked to rate their pain on the study-specific Lingard pain scale post-cystocopy.
  The Lingard pain scale is an outcome measure scaled from 0 (no pain) to 10 (pain as bad it could be). The higher the reported rating out of 10, the more pain the participant has experienced.

CONTACTS AND LOCATIONS:
Locations (1):
- Heidi Wagner, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No